CLINICAL TRIAL: NCT01225276
Title: Double-blind, Placebo-controlled, Randomised, Multicentre, Adaptive, Two-stage Phase 2/3 Study Evaluating Safety and Efficacy of Three Dosages of NewGam in CIDP Patients
Brief Title: Safety and Efficacy Study of Three Different Dosages of NewGam in Patients With CIDP
Acronym: POINT
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Study Terminated.priority changes in product development.
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NGAM-03
Record Dates: First submitted 2010-10-06; First posted 2010-10-20 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Chronic Inflammatory Demyelinating Polyradiculoneuropathy
Keywords: CIDP; IVIG
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Dosage Arm 1 (Experimental): NewGam 10% 0.4 g/kg
  Interventions: Drug: NewGam 10%
- Dosage Arm 2 (Experimental): NewGam 10% 1.0 g/kg
  Interventions: Drug: NewGam 10%
- Dosage Arm 3 (Experimental): NewGam 10% 2.0 g/kg
  Interventions: Drug: NewGam 10%
- Dosage Arm 4 (Placebo Comparator): Placebo 0.9% Saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NewGam 10% — Loading dose at baseline (Week 0) will be 2.0 g/kg NewGam . The maintenance doses to be infused 7 times will be 2.0 g/kg every 21 (+/-4) days.
  Arms: Dosage Arm 1
Drug: Placebo — Loading dose at baseline (Week 0) in Placebo arm will be corresponding volume of an authorised 0.9% saline solution . The maintenance doses of the 0.9% saline solution to be infused 7 times will be given every 21 (+/-4) days.
  Other Names: 0.9% saline solution
  Arms: Dosage Arm 4
Drug: NewGam 10% — Loading dose at baseline (Week 0) will be 2.0 g/kg NewGam in all three NewGam treatment arms. The maintenance doses to be infused 7 times will be 1.0 g/kg every 21 (+/-4) days.
  Arms: Dosage Arm 2
Drug: NewGam 10% — Loading dose at baseline (Week 0) will be 2.0 g/kg NewGam in all three NewGam treatment arms. The maintenance doses to be infused 7 times will be 0.4 g/kg every 21 (+/-4) days.
  Arms: Dosage Arm 3

SUMMARY:
NewGam (current working title for a new IGIV formulation) is a newly developed human normal immunoglobulin solution ready for intravenous administration (IGIV). This study will evaluate the safety and efficacy of three different dosages of NewGam 10% in patients with Chronic Inflammatory Demyelinating Polyradiculoneuropathy.

DETAILED DESCRIPTION:
This is a Phase 2/3 study that will take place in 2 stages. The primary objective of Stage 1 (Phase 2 dose-finding part)is to determine and select one dosage from three NewGam maintenance dosage arms in comparison with a placebo arm, based on the percentage of responders (response defined as a decrease, meaning improvement, in the adjusted INCAT disability score by at least 1 point). The selected NewGam dosage and placebo will be employed and compared in Stage 2.

The primary objective of Stage 2 (Phase 3 confirmatory part) is to demonstrate superiority of the maintenance dosage regimen selected at study Stage 1 over placebo in patients with CIDP as assessed by the percentage of responders.

The secondary objective is to evaluate the safety (measured by number of adverse events)and efficacy of NewGam administration in patients with CIDP compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as having CIDP based on fulfilment of clinical criteria of the INCAT Group and the definite electrophysiological criteria for CIDP ; patients with MADSAM or pure motor CIDP will be included provided they fulfil these criteria
* Worsening of disability and objective increase in weakness or sensory deficit during the 6 months prior to screening
* >=18 years of age

Exclusion Criteria:

* Unifocal forms of CIDP
* Pure sensory CIDP
* MMN with conduction block
* Treatment of CIDP with immunoglobulins (intravenous or subcutaneous) at any time prior to study entry
* Steroids of any type equivalent to prednisolone or prednisone > 10 mg/day or equivalent plasma exchange (PE) during the last 3 months prior to baseline visit
* Treatment with cyclosporin, methotrexate, mitoxantrone, mycophenolate mofetil, interferon or other immunosuppressive or immunomodulatory drugs during the three months prior to baseline visit
* Clinical evidence of peripheral neuropathy from another
* Known diabetes mellitus
* Other serious medical condition complicating assessment or treatment
* Thromboembolic events: patients with a history of deep vein thrombosis (DVT) within the last year prior to baseline visit or pulmonary embolism ever
* Known IgA deficiency with antibodies to IgA
* History of hypersensitivity, anaphylaxis or severe systemic response to immunoglobulin, blood or plasma derived products, or any component of NewGam
* Known blood hyperviscosity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Adjusted INCAT disability score | Every 3 weeks for 48 weeks (stage 1) or 36 weeks (stage 2)

SECONDARY OUTCOMES:
Vital Signs | During each infusion - Every 3 weeks for 48 weeks (stage 1) or 36 weeks (stage 2)
Grip Strength | Visit 9 & 13
Nerve Conduction Studies | Visti 9 & 13
Motor Impairment Assessment utlizing the Expanded MRC Sum Score | Every 3 weeks for 48 weeks (stage 1) or 36 weeks (stage 2)
  Expanded 'Medical Research Council sum score' will be measured as improvement in MRC units .

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Frenzel, MD, Study Director — Octapharma

IPD SHARING:
Plan to Share IPD: No
no (IPD) data exist for this study

REFERENCES:
- [Derived] Bus SR, de Haan RJ, Vermeulen M, van Schaik IN, Eftimov F. Intravenous immunoglobulin for chronic inflammatory demyelinating polyradiculoneuropathy. Cochrane Database Syst Rev. 2024 Feb 14;2(2):CD001797. doi: 10.1002/14651858.CD001797.pub4. PMID 38353301